CLINICAL TRIAL: NCT04277585
Title: Improving Access to Early Psychosis Coordinated Specialty Care Services
Brief Title: Improving Access to Early Psychosis Coordinated Specialty Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0048; 3B09SM010032-19S3 (SAMHSA)
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Psychosis
Keywords: Telehealth; Specialty Care; Rural Initiative
MeSH Terms: conditions — Psychotic Disorders | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Open feasibility trial of addition of telehealth to an Early Psychosis Coordinated Specialty Service
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OASIS Clients (Experimental): Clients of the OASIS Program who live at least 45 minutes away from an Early Psychosis Coordinated Specialty Care Program and are willing to engage in some of their services through telehealth.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — Early Psychosis Coordinated Specialty Care Services via telehealth.
  Other Names: Video visits

SUMMARY:
The aim of this study is to evaluate the feasibility of developing an Early Psychosis CSC service delivery model suitable for rural settings in NC. Major challenges to delivery of specialized health care services for persons in the early stages of psychosis include the high level of provider expertise and the frequency and intensity of services. These challenges limit the feasibility of brick-and-mortar programs to serve individuals living in rural settings. This study proposes to expand service delivery methods to include telehealth as a potential solution.

DETAILED DESCRIPTION:
The UNC OASIS program currently provides evidenced-based outpatient coordinated specialty care services (CSC) to persons within the first five years of a psychotic disorder. Medical management and psychotherapy services are mainly provided in brick and mortar offices. Supported education, supported employment, and peer support services are provided in offices and also in the community. The service model is relatively intense, involving treatment sessions up to several times a week. Thus a barrier to persons in rural North Carolina receiving CSC services is the time taken to travel to office based appointments.

The purpose of this study is to determine feasibility and acceptability of providing some of the services provided by OASIS via telehealth.

Participants: Up to 10 patients who have been accepted by the OASIS program and who live 45-minutes or more from the UNC OASIS program or another CSC program. Participants must also have home internet bandwidth sufficient to support the telehealth platform and own a computer or other device (smart phone, tablet, etc.) compatible with the telehealth platform.

Procedures (methods): The OASIS program does not exclude patients based on where they live in North Carolina. Potential OASIS patients and their families participate in an initial psychosocial and medical evaluation. At this time the OASIS program director reviews the OASIS program expectations with the patient and family. If the OASIS program and the patient and the patient's family member agree that the OASIS program is a good fit, the patient is then accepted into the program. After acceptance into the OASIS program patients who live 45 minutes or more away from the UNC OASIS or another CSC program and who reside in North Carolina will be informed about the availability of the telehealth pilot project by the OASIS program director.

UNCH has developed a telehealth service that is provided via the UNC electronic medical record platform, EPIC. If interested, the OASIS patient and their family member will meet with a study staff person, who will evaluate whether their internet bandwidth is sufficient to support the EPIC telehealth platform and if they own a computer or other device that supports the EPIC telehealth platform. Patients who are interested and who meet these requirements will then participate in the oral and written informed consent process.

Participants who consent to participate in the study will receive some of their CSC services via telehealth, and will continue to receive some of their services in the OASIS offices. During this pilot phase the project will be flexible about the relative proportion of services delivered via telehealth and in-person. The main study participant is the patient, however since family therapy may be delivered via telehealth interested family members are also asked to consent to study participation.

The OASIS program routinely collects quality assurance data via self-report and clinician-administered assessments. The study will obtain consent from study participants to access this information. In addition to the Quality Assurance document patients who are subjects and their family members who also consent to participate in the the telehealth pilot project will also complete a self-report survey inquiring about their satisfaction with telehealth services.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-36
* Reside in NC
* Live more than a 45 minute drive from UNC OASIS or UNC Encompass CSC programs.
* Accepted into the OASIS program.
* Have access to a computer or other device with broadband internet sufficient to support the EPIC-delivered telehealth services.
* Willing to receive some services via telehealth. A family member of a patient who is participating in this research study.

Exclusion Criteria:

* Not age 18-36
* Does not reside in NC
* Live within a 45 minute drive from UNC OASIS or UNC Encompass CSC programs.
* Not accepted into the OASIS program.
* No access to a computer or other device with broadband internet sufficient to support the EPIC-delivered telehealth services.
* Not willing to receive any services via telehealth

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Mean Telehealth Healthcare Service Satisfaction and Usability Score (Month 3) | 3 months
  The UNC OASIS Telehealth Satisfaction and Usability Survey is a self-report measure with 8 items assessing satisfaction with aspects of telehealth service delivery. Items using 5-item likert scale ranged from Strongly agree to Strongly disagree. Items include: 1) sessions ran smoothly, 2) preference for in-person or telehealth service or no preference, 3) comfortable using telehealth technology, 4) technical difficulties encountered (5-item likert ranging from Never to Often), 5) privacy/confidentiality of telehealth as either better than/same as/not as good as in-person visits and any comments, 6) comfort level communicating to staff using telehealth, 7) whether telehealth made attending appointments easier/same as/more difficult than in person visits, 8) whether would use telehealth services again. Lower scores reflect higher satisfaction.
Mean Telehealth Healthcare Service Satisfaction and Usability Score (Month 6) | 6 months
  The UNC OASIS Telehealth Satisfaction and Usability Survey is a self-report measure with 8 items assessing satisfaction with aspects of telehealth service delivery. Items using 5-item likert scale ranged from Strongly agree to Strongly disagree. Items include: 1) sessions ran smoothly, 2) preference for in-person or telehealth service or no preference, 3) comfortable using telehealth technology, 4) technical difficulties encountered (5-item likert ranging from Never to Often), 5) privacy/confidentiality of telehealth as either better than/same as/not as good as in-person visits and any comments, 6) comfort level communicating to staff using telehealth, 7) whether telehealth made attending appointments easier/same as/more difficult than in person visits, 8) whether would use telehealth services again. Lower scores reflect higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Perkins, MD, MPH, Principal Investigator — University of North Carolina, School of Medicine, Department of Psychiatry
Locations (1):
- OASIS Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: 9-36 months following publication
Access Criteria: IRB/IEC/REB approval and executed data use/sharing agreement with UNC.